CLINICAL TRIAL: NCT07255079
Title: A Randomized, Blinded, Comparator Controlled, Cross-over Clinical Trial to Assess the Pharmacokinetic Profile of Three Coenzyme Q10 Formulations in Healthy Adults
Brief Title: A Clinical Trial to Assess the Pharmacokinetic Profile of Three Coenzyme Q10 Formulations in Healthy Adults
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: 3i Solutions (Industry)
Collaborators: KGK Science Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Other
Other Study IDs: 25IIIRR01
Record Dates: First submitted 2025-11-20; First posted 2025-11-28 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Pharmacokinetic Parameters; Bioavailability Heathy Volunteers
Keywords: pharmacokinetic; bioavailability; healthy volunteers; Coenzyme Q10
MeSH Terms: interventions — coenzyme Q10

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- VitaDry-CoQ10 (Experimental): VitaDry CoQ10 contains 100 mg of CoQ10 per serving.
  Interventions: Dietary Supplement: VitaDry-Q10
- VitaSperse-CoQ10 (Experimental): VitaSperse-CoQ10 contains 50 mg of CoQ10 per serving.
  Interventions: Dietary Supplement: VitaSperse-Q10
- CoQ10 (Experimental): CoQ10 contains 50 mg of CoQ10 mg per serving.
  Interventions: Dietary Supplement: Coenzyme Q10

INTERVENTIONS:
Dietary Supplement: VitaDry-Q10 — Participants consuming a capsule product will be required to consume 2 x 50mg capsules for a combined dose of 100mg with a cup of water.
  Arms: VitaDry-CoQ10
Dietary Supplement: VitaSperse-Q10 — Participants consuming liquid product will be required to drink a cup of water following administration of 5 mL of study product delivered via syringe.
  Arms: VitaSperse-CoQ10
Dietary Supplement: Coenzyme Q10 — Participants consuming a capsule product will be required to consume 2 x 50mg capsules for a combined dose of 100mg with a cup of water.
  Arms: CoQ10

SUMMARY:
The goal of this clinical trial is to assess the pharmacokinetic profile of three Coenzyme Q10 formulations in healthy adults. The main question it aims to answer is:

What is the difference in the bioavailability of three Coenzyme Q10 (CoQ10) formulations as assessed by the incremental area-under-the-curve (AUC) from time 0 to the last measured timepoint (AUC0-72hr)?

Participants will be asked to consume three formulations of CoQ10 and will be evaluated for CoQ10 levels in blood, over a 71-day period.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females ≥ 18 years of age
2. BMI between 18.5 to 29.9 Kg/m3, inclusive
3. Females not of child-bearing potential, defined as those who have undergone a sterilization procedure (e.g. hysterectomy, bilateral oophorectomy, bilateral tubal ligation, complete endometrial ablation) or have been post-menopausal for at least 1 year prior to screening

   Or,

   Individuals of child-bearing potential must have a negative baseline urine pregnancy test and agree to use a medically approved method of birth control for the duration of the study. All hormonal birth control must have been in use for a minimum of three months. Acceptable methods of birth control include:
   * Hormonal contraceptives including oral contraceptives, hormone birth control patch (Ortho Evra), vaginal contraceptive ring (NuvaRing), injectable contraceptives (Depo-Provera, Lunelle), or hormone implant (Norplant System)
   * Double-barrier method
   * Intrauterine devices
   * Non-heterosexual lifestyle and agrees to use contraception if planning on changing to heterosexual partner(s)
   * Vasectomy of partner at least 6 months prior to screening
   * Abstinence and agrees to use contraception if planning on becoming sexually active during the study
4. Willingness to complete questionnaires and diaries associated with the study and complete all study requirements
5. Agrees to maintain current lifestyle (diet, physical activity, medications, supplements, and sleep) as much as possible within study specific requirements throughout the study
6. Provided voluntary, written, informed consent to participate in the study
7. Healthy as determined by medical history and laboratory results as assessed by the Qualified Investigator (QI)

Exclusion Criteria:

1. Individuals who are pregnant, breast feeding, or planning to become pregnant during the study
2. Poor venous access, as assessed by the QI
3. Allergy, sensitivity, intolerance, or dietary restriction preventing consumption of investigational products or comparator ingredients or inability to consume the standardized meals
4. Following a specific diet (e.g. vegetarian, carnivore, paleo, vegan, etc.…)
5. Unstable metabolic disease or chronic diseases as assessed by the QI
6. Current or history of any significant diseases of the gastrointestinal tract as assessed by the QI
7. Unstable hypertension. Treatment on a stable dose of medication for at least 3 months will be considered by the QI
8. Type I or Type II diabetes
9. Significant cardiovascular event in the past 6 months. Participants with no significant cardiovascular event on stable medication may be included after assessment by the QI on a case-by-case basis
10. History of or current diagnosis with kidney and/or liver diseases as assessed by the QI on a case-by-case basis, with the exception of history of kidney stones in participants who are symptom free for 6 months
11. Self-reported confirmation of current or pre-existing thyroid condition. Treatment on a stable dose of medication for at least 3 months will be considered by the QI
12. Major surgery in the past 3 months or individuals who have planned surgery during the course of the study. Participants with minor surgery will be considered on a case-by-case basis by the QI
13. Cancer, except skin basal cell carcinoma completely excised with no chemotherapy or radiation with a follow up that is negative. Volunteers with cancer in full remission for more than five years after diagnosis are acceptable
14. Individuals with an autoimmune disease or are immune compromised as assessed by the QI
15. Self-reported confirmation of a HIV-, Hepatitis B- and/or C-positive diagnosis as assessed by the QI
16. Self-reported confirmation of blood/bleeding disorders as assessed by the QI
17. Use of medical cannabinoid products
18. Chronic use of cannabinoid products (>2 times/week). Occasional users will be required to washout and abstain for the duration of the study period
19. Regular use of tobacco or nicotine products in the past six months, as assessed by the QI. Occasional users will be required to washout and abstain for the duration of the study period
20. Alcohol intake average of >2 standard drinks per day as assessed by the QI
21. Alcohol or drug abuse within the last 12 months
22. Current use of prescribed and/or over-the-counter (OTC) medications, supplements, and/or consumption of food/drinks that may impact the efficacy and/or safety of the investigational product (Sections 7.3.1 and 7.3.2)
23. Clinically significant abnormal laboratory results at screening as assessed by the QI
24. Blood donation 30 days prior to baseline, during the study, or a planned donation within 30 days of the last study visit
25. Participation in other clinical research studies 30 days prior to baseline, as assessed by the QI
26. Individuals who are unable to give informed consent
27. Any other condition or lifestyle factor, that, in the opinion of the QI, may adversely affect the participant's ability to complete the study or its measures or pose significant risk to the participant

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Difference in the bioavailability of three Coenzyme Q10 (CoQ10) formulations as assessed by the incremental area-under-the-curve (AUC) | 0 to 72 hours post dose
  Difference in the bioavailability of three Coenzyme Q10 (CoQ10) formulations as assessed by the incremental area-under-the-curve (AUC) from time 0 to the last measured timepoint (AUC0-72hr)

SECONDARY OUTCOMES:
Difference in incremental AUC between three CoQ10 formulations | 0 hours to infinity post dose
  Difference in incremental AUC between three CoQ10 formulations from time 0 to infinity (AUC0-∞)
Difference in AUC between three CoQ10 formulations | 0 hours to 72 hours post dose
  Difference in AUC between three CoQ10 formulations from time 0 to 72 hours (AUC0-72hr)
Difference in Maximum concentration (Cmax) between three CoQ10 formulations | 0 hours to Cmax post dose
  Difference in Maximum concentration (Cmax) between three CoQ10 formulations
Difference in time to peak maximum concentration (tmax) between three CoQ10 formulations | 0 hours to tmax post dose
  Difference in time to peak maximum concentration (tmax) between three CoQ10 formulations
Difference in half-life (t1/2) between three CoQ10 formulations | 0 hours to tmax post dose
  Difference in half-life (t1/2) between three CoQ10 formulations

OTHER OUTCOMES:
Clinically relevant changes in heart rate after supplementation. | Day 0 to 71
  Clinically relevant changes in heart rate after supplementation. Safety outcome where clinically relevant changes refer to the opinion of the Qualified Investigator that changes indicates there is an Adverse Event.
Clinically relevant changes in blood pressure (BP) after supplementation | Day 0 to 71
  Clinically relevant changes in heart rate after supplementation. Safety outcome where clinically relevant changes refer to the opinion of the Qualified Investigator that changes indicates there is an Adverse Event.
Incidence of post-emergent adverse events (AE) | Day 0 to 71
  Incidence of post-emergent adverse events (AE)
Clinically relevant changes in complete blood count after supplementation | Day 0 to 71
  Clinically relevant changes in complete blood count after supplementation

CONTACTS AND LOCATIONS:
Locations (1):
- KGK Science Inc., London, Ontario, Canada